CLINICAL TRIAL: NCT04327401
Title: COVID-19-associated ARDS Treated With DEXamethasone: an Open-label, Randomized, Controlled Trial: CoDEX (Alliance Covid-19 Brasil III)
Brief Title: COVID-19-associated ARDS Treated With Dexamethasone: Alliance Covid-19 Brasil III
Acronym: CoDEX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Data Monitoring Committee recommended to stop the trial based on the Recovery Trial results, which was accepted by the CoDEX Steering Committee.
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: Hospital Israelita Albert Einstein (Other); Hospital do Coracao (Other); Brazilian Research In Intensive Care Network (Network); Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Principal Investigator, Luciano Cesar Pontes de Azevedo, Research Director, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 30227020.5.1001.0008
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Coronavirus Infection; Pneumonia, Viral; Acute Respiratory Distress Syndrome
Keywords: SARS-CoV2 virus; 2019-nCOV; Dexamethasone; ARDS; Corticosteroids; Respiratory failure
MeSH Terms: conditions — Coronavirus Infections; Pneumonia, Viral; Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: 1. Dexamethasone. After randomization, dexamethasone 20mg IV 1x/day for 5 days, followed by 10mg IV 1xd for 5 days + standard treatment (according to the treatment protocol for 2019-nCoV infection).
  2. Standard treatment (according to the treatment protocol for 2019-nCoV infection).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Dexamethasone. After randomization, dexamethasone [20mg IV 1x/day for 5 days, followed by 10mg IV 1xd for 5 days] + standard treatment (according to the treatment protocol for 2019-nCoV infection).
  Interventions: Drug: Dexamethasone
- Control (No Intervention): Standard treatment (according to the treatment protocol for 2019-nCoV infection).

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone administration for 10 consecutive days after randomization.
  Other Names: Decadron; Dexasone; Diodex; Hexadrol; Maxidex
  Arms: Intervention group

SUMMARY:
The Severe Acute Respiratory Syndrome COronaVirus 2 (SARS-CoV2) is a new and recognized infectious disease of the respiratory tract. Most cases are mild or asymptomatic. However, around 5% of all patients develop Acute Respiratory Distress Syndrome (ARDS), which is the leading mortality cause in these patients. Corticosteroids have been tested in deferent scenarios of ARDS, including viral pneumonia, and the early use of dexamethasone is safe and appears to reduce the duration of mechanical ventilation in ARDS patients. Nevertheless, no large, randomized, controlled trial was performed evaluating the role of corticosteroids in patients with ARDS due SARS-CoV2 virus. Therefore, the present study will evaluate the effectiveness of dexamethasone compared to control (no corticosteroids) in patients with moderate and severe ARDS due to SARS-CoV2 virus.

DETAILED DESCRIPTION:
The Severe Acute Respiratory Syndrome COronaVirus 2 (SARS-CoV2) is a new and recognized infectious disease of the respiratory tract, and its outbreak deemed a pandemic in early March 2020. Estimates show around 5% of all patients develop Acute Respiratory Distress Syndrome (ARDS), which due to its severity, consumes most Intensive Care Units (ICU) resources and is the leading mortality cause in this population. Given its burden, therapies that reduce the duration of mechanical ventilation or decrease the morbimortality are needed. Studies indicate that inflammation and cytokine storm might be involved in the pathophysiological pathway to ARDS in these patients. Corticosteroids have been tested in deferent scenarios of ARDS, including viral pneumonia, and the early use of dexamethasone is safe and appears to reduce the duration of mechanical ventilation in ARDS patients. A recent small retrospective study evaluating the role of corticosteroids found no association between corticosteroids and hospital length of stay, virus clearance, and symptoms' duration. However, the retrospective nature of data, small sample size (31 patients), and no protocol for corticosteroids administration undermine its results. Therefore, the present study will evaluate the effectiveness of dexamethasone compared to control (no corticosteroids) in ventilator-free days at 28 days in patients with moderate and severe ARDS due to SARS-CoV2 virus in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Probable or confirmed infection by SARS-CoV2
* Intubated and mechanically ventilated
* Moderate/severe ARDS defined by the Berlin criteria (PaO2/FiO2 ≤200mmHg with PEEP ≥5cmH20)
* Onset of moderate/severe ARDS in less than 48 hours before randomization

Exclusion Criteria:

* Pregnancy or active lactation
* Known history of dexamethasone allergy
* Daily use of corticosteroids in the past 15 days
* Clinical indication for corticosteroids use for other diseases (i.e refractory septic shock)
* Patients who did use corticosteroids during hospital stay for periods equal or greater than two days
* Use of immunosuppressive drugs
* Cytotoxic chemotherapy in the past 21 days
* Neutropenia due to hematological or solid malignancies with bone marrow invasion
* Patient expected to die in the next 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days | 28 days after randomization
  Ventilator-free days, defined as alive and free from mechanical ventilation, at 28 days after randomization.

SECONDARY OUTCOMES:
Evaluation of the clinical status | 15 days after randomization
  Evaluation of the clinical status of patients on the 15th day after randomization defined by the 6-point Ordinal Scale, this scale ranges from 1 (Not hospitalized) to 6 (Death) with higher scores meaning worse outcomes.
All-cause mortality | 28 days after randomization
  All-cause mortality rates at 28 days after randomization.
Mechanical ventilation duration | 28 days after randomization
  Number of days of mechanical ventilation from randomization to day 28.
Sequential Organ Failure Assessment (SOFA) Score | Score at 48 hours, 72 hours and 7 days after randomization
  Sequential Organ Failure Assessment (SOFA) Score 48 hours, 72 hours and 7 days after randomization

OTHER OUTCOMES:
Intensive Care Unit free days | 28 days after randomization
  Intensive Care Unit free days, defined as alive and discharged from the intensive care unit, at 28 days after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Cesar Pontes Azevedo, Ph.D, Principal Investigator — Teaching Director of Teaching & Research Institute Sírio-Libanês Hospital
Locations (21):
- Brazil (21):
  - Fundação Social Rural de Colatina, Colatina, Esoírito Santo
  - Hospital Ana Nery, Salvador, Estado de Bahia
  - Instituto de Cardiologia do Distrito Federal, Brasília, Federal District
  - Hospital Vera Cruz AS, Belo Horizonte, Minas Gerais
  - Hospital Maternidade E Pronto Socorro Santa Lucia Ltda, Poços de Caldas, Minas Gerais
  - Universidade Estadual de Londrina, Londrina, Paraná
  - Eurolatino Natal Pesquisas Médicas Ltda, Natal, Rio Grande do Norte
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Maestri E Kormann Consultoria Medico-Cientifica, Blumenau, Santa Catarina
  - Sociedade Literaria e Caritativa Santo Agostinho, Criciúma, Santa Catarina
  - Fundação Pio XII, Barretos, São Paulo
  - Santa Casa de Misericordia de Votuporanga, Votuporanga, São Paulo
  - Associacao Beneficente Siria, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da USP - HCFMRP, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Prevent Senior Private Operadora de Saude Ltda, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência/SP, São Paulo
  - Santa Casa de Misericórdia, São Paulo
  - Secretaria de Saúde do Estado de São Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sírio-Libanês, São Paulo
  - Universidade Federal de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tomazini BM, Maia IS, Cavalcanti AB, Berwanger O, Rosa RG, Veiga VC, Avezum A, Lopes RD, Bueno FR, Silva MVAO, Baldassare FP, Costa ELV, Moura RAB, Honorato MO, Costa AN, Damiani LP, Lisboa T, Kawano-Dourado L, Zampieri FG, Olivato GB, Righy C, Amendola CP, Roepke RML, Freitas DHM, Forte DN, Freitas FGR, Fernandes CCF, Melro LMG, Junior GFS, Morais DC, Zung S, Machado FR, Azevedo LCP; COALITION COVID-19 Brazil III Investigators. Effect of Dexamethasone on Days Alive and Ventilator-Free in Patients With Moderate or Severe Acute Respiratory Distress Syndrome and COVID-19: The CoDEX Randomized Clinical Trial. JAMA. 2020 Oct 6;324(13):1307-1316. doi: 10.1001/jama.2020.17021. PMID 32876695

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT04327401/Prot_SAP_000.pdf